CLINICAL TRIAL: NCT00726271
Title: A Pilot 6 Week Study of the Feasibility and Acceptability of Dietary Modification With the Goal of Changing the Appetite Set Point in People Taking Medications That Cause Weight Gain Through Increased Appetite.
Brief Title: Pilot Study of Dietary Modification of Appetite Set Point in Obesity
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Record owner left institution
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Lisa Kaufmann, MD, SUNY Upstate Medical University, Syracuse, NY 13210
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5653
Record Dates: First submitted 2008-07-28; First posted 2008-07-31 (Estimated); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Obesity
Keywords: obesity; appetite set point
MeSH Terms: conditions — Obesity | interventions — Linseed Oil; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- active (Experimental): Subjects will complete the Zung Depression and Anxiety Scales. At the first visit the subject's medication list, weight, height, and waist measurement will be obtained. The goal is to recruit a minimum of 20 patients.
  Subjects will receive light olive oil, and capsules of fish oil and flaxseed oil, to take daily at home with weight based dosing, based on the doses recommended in Dr. Roberts' work. Doses are within the recommended dietary ranges to improve intermediate outcomes for coronary artery disease subjects.
  They will return weekly for measurement of weight, waist measurements, discussion of any problems with the oils, and dose adjustment of the oils.
  Interventions: Dietary Supplement: light olive oil, fish oil capsules, flax seed oil capsules

INTERVENTIONS:
Dietary Supplement: light olive oil, fish oil capsules, flax seed oil capsules — fish oil 1000 mg capsules three daily flax seed oil 1000 mg capsules three daily light olive oil 30 ml to 60 ml daily(weight less than 160 pounds, 30 ml/ weight 160-200 pounds 45 ml/ weight over 200 pounds 60 ml)
  Other Names: Naturemade brand flax seed and fish oils; Wegman's store brand light olive oil

SUMMARY:
An innovative dietary approach to obesity, based on the set-point theory of body weight and associative learning, was developed by Seth Roberts. Roberts's approach focuses on dissociating flavor and calories by consuming small amounts of very bland but calorie-dense foods such as extra-light olive oil between meals. Roberts believes that the dissociation between flavor and calories lowers the body weight's set point, suppressing appetite and thereby inducing weight loss without causing hunger. Studying the feasibility of this approach is particularly relevant to patients taking drugs that cause increased appetite and weight gain as a side effect, as increased hunger makes the usual calorie restriction approach even more difficult than it normally is. Low-income people have a diet higher in prepackaged standardized foods, which may be one contributing factor to their higher risk of developing obesity.

Specific Aims

* To test the acceptance of, and the patients' compliance rate to, the Shangri-La Diet
* To ascertain whether a controlled clinical trial of the Shangri-La Diet would be feasible.
* To see if the weight loss documented anecdotally in many people is reproducible in patients from low-income areas who are overweight and taking prescribed medications associated with increased appetite and weight gain.

Analysis: The primary end point will be acceptability of the dietary intervention as measured by the final interview and the evaluation form-is this something patients would be willing to do over the long term? This will help determine whether a controlled trial of the dietary intervention would be feasible, and provide information needed to design such a trial. Secondary outcomes will be changes in the participants' weight, waist measurements, anxiety, and depression scores

DETAILED DESCRIPTION:
An innovative dietary approach to obesity, based on the set-point theory of body weight and associative learning, was developed by Seth Roberts, professor of psychology at the University of California at Berkeley. The set-point theory was first proposed by G. Kennedy, who hypothesized that body fat, like body temperature, is controlled by a set point in a thermostat-like system. Based on this theory and subsequent work, Roberts hypothesized that people have a strong conditioned response to specific food items, which raises the weight set point, like a thermostat, stimulating appetite and storing the excess calories as fat. In an environment with attractive, easily accessible, inexpensive food, many people will gain weight. Roberts also hypothesizes that consistency in the presentation, labeling, and taste of mass produced food items today elicits a stronger conditioned response than in the past. Roberts's approach focuses on dissociating flavor and calories by consuming small amounts of very bland but calorie-dense foods such as extra-light olive oil or sugar water between meals. Roberts believes that the dissociation between flavor and calories lowers the body weight's set point, suppressing appetite and thereby inducing weight loss without causing hunger. Decreased oral intake naturally follows a decrease in appetite, without the hunger that normally quickly appears when people reduce their caloric intake, so people can eat an amount that feels comfortable without conscious dietary restriction. Roberts outlined this approach in a book titled "The Shangri-La Diet" because it is not really a diet at all. Given the originality of this approach, the successful outcomes accounted in the book and in anecdotes on the internet definitely warrant a closer look. Studying the feasibility of the Shangri-La Diet is particularly relevant to patients taking drugs that cause increased appetite and weight gain as a side effect, as increased hunger makes the usual calorie restriction approach even more difficult than it normally is. Low-income people have a diet higher in prepackaged standardized foods, which may be one contributing factor to their higher risk of developing obesity.

Specific Aims

* To test the acceptance of, and the patients' compliance rate to, the Shangri-La Diet
* To ascertain whether a controlled clinical trial of the Shangri-La Diet would be feasible.
* To see if the weight loss documented anecdotally in many people is reproducible in patients from low-income areas who are overweight and taking prescribed medications associated with increased appetite and weight gain.

Methods

2. Subjects will receive light olive oil, and capsules of fish oil and flaxseed oil, to take daily at home with weight based dosing, based on the doses recommended in Dr. Roberts' work. Doses are within the recommended dietary ranges to improve intermediate outcomes for coronary artery disease (HDL, LDL, and triglycerides) and ranges associated with a decreased risk of cardiac and all cause mortality in epidemiological studies. They will return weekly for measurement of weight, waist measurements, discussion of any problems with the oils, and dose adjustment of the oils.

3. Evaluation: At the end of 6 weeks of the intervention, the subjects will complete the same questionnaires as at baseline, and an evaluation form about the intervention.

Analysis: The primary end point will be acceptability of the dietary intervention as measured by the final interview and the evaluation form-is this something patients would be willing to do over the long term? Secondary outcomes will be changes in the participants' weight, waist measurements, anxiety, and depression scores.

ELIGIBILITY:
Inclusion Criteria:

1. Must be taking at least one medication that is described in the Lexi-comp data base used by SUNY Upstate Medical University Hospital for drug information, as potentially causing weight gain
2. BMI must be over 29
3. Must be fluent in English
4. Must have access to a telephone
5. Must be able and willing to come in for weekly measurements during the six weeks
6. Must not be known to be currently hypothyroid or hyperthyroid. Someone who is euthyroid on replacement could be eligible

Exclusion Criteria:

1. Inability to fully understand the protocol and consent form, including people who have active psychosis
2. Type 1 Diabetes
3. Inability to read at the 4th grade level
4. Current alcohol abuse as determined by the primary provider, or illicit substance use
5. Current warfarin use
6. Bleeding disorder or thrombocytopenia
7. Allergy to fish oil, flaxseed oil, or olive oil
8. Current use of any medication that has a probable negative interaction with any of the oils used in the intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
acceptability and adherence to the dietary intervention | 6 weeks

SECONDARY OUTCOMES:
weight | 6 weeks
waist circumference | 6 weeks
body mass index | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Kaufmann, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States